CLINICAL TRIAL: NCT05943639
Title: The Effect of Cultural Marginality Theory-Based Education on Intercultural Adaptation and Psychological Well-Being of Foreign Nursing Students: A Randomized Controlled Study
Brief Title: Effect of Cultural Marginality Theory-Based Education on Intercultural Adaptation and Psychological Well-Being of Foreign Nursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hilal Altundal (Other)
Responsible Party: Sponsor-Investigator, Hilal Altundal, Doctor, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ÇankırıKaratekinU
Record Dates: First submitted 2023-06-26; First posted 2023-07-13 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Culture; Adaptation, Psychological; Psychological Well-being
Keywords: randomized controlled trial; foreign nursing student; psychological well-being; intercultural adaptation; cultural marginality
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study was planned as a prospective, two-armed (1:1), randomized controlled experimental study. This randomized controlled trial will be reported according to the CONSORT guidelines.
Who Masked: Participant
Masking Description: Foreign students in the experimental and control groups will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The Cultural Marginality Theory-Based Education program will be held in a face-to-face classroom environment for the students in the experimental group. This training program has been developed based on the concepts of Cultural Marginality Theory. The content and topics of the sessions in the program are arranged according to the conceptual structure and flow of the theory. The training program was created in a certain flow, based on the concepts of recognizing intercultural conflict (2 sessions), marginal living (2 sessions) and alleviating cultural tension (2 sessions). There are 6 sessions in the program and the frequency of sessions is 2 times a week, and each session lasts approximately 45 minutes. The training program will be applied to 33 foreign nursing students in the experimental group.
  Interventions: Other: The Cultural Marginality Theory-Based Education
- Control group (No Intervention): There will be no training or intervention.

INTERVENTIONS:
Other: The Cultural Marginality Theory-Based Education — The Cultural Marginality Theory-Based Education program will be held in a face-to-face classroom environment for the students in the experimental group. This training program has been developed based on the concepts of Cultural Marginality Theory. The content and topics of the sessions in the program are arranged according to the conceptual structure and flow of the theory. The training program was created in a certain flow, based on the concepts of recognizing intercultural conflict (2 sessions), marginal living (2 sessions) and alleviating cultural tension (2 sessions). There are 6 sessions in the program and the frequency of sessions is 2 times a week, and each session lasts approximately 45 minutes. The training program will be applied to 33 foreign nursing students in the experimental group.
  Arms: Experimental group

SUMMARY:
In this study, between 1 - 31 December 2022, who met the inclusion and exclusion criteria, a total of 66 foreign nursing students who are with 1st year foreign students starting the Nursing Department of Ondokuz Mayıs University and Mersin University.

DETAILED DESCRIPTION:
The Cultural Marginality Theory-Based Education program will be held in a face-to-face classroom environment for the students in the experimental group. This training program has been developed based on the concepts of Cultural Marginality Theory. The content and topics of the sessions in the program are arranged according to the conceptual structure and flow of the theory. The training program was created in a certain flow, based on the concepts of recognizing intercultural conflict (2 sessions), marginal living (2 sessions) and alleviating cultural tension (2 sessions). There are 6 sessions in the program and the frequency of sessions is 2 times a week, and each session lasts approximately 45 minutes. The training program will be applied to 33 foreign nursing students in the experimental group. In the first session to the students in the experimental group and to the students in the control group after the post-tests, the training booklet, which consists of information about the educational content in the program, will be given online in pdf format in color and with pictures.

ELIGIBILITY:
Inclusion Criteria:

1. being a first-year foreign nursing student studying at state universities in the north and south two cities of Türkiye,
2. agreeing to participate in the research
3. not having communication barrier

Exclusion Criteria:

1) having a physical or mental illness that would prevent participation in the research

The Termination Criteria:

1. withdrawing from the research voluntarily
2. not attending at least one of the sessions
3. incomplete or incorrectly answering the instruments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-09-15 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
CROSS CULTURAL ADAPTABILITY INVENTORY (CCAI) | Change from before education up to after education (three weeks)
  The Turkish adaptation of the inventory developed by Kelley and Meyers in 1992 was made in 2009 by Karaeminoğulları, Doğan and Bozkurt. The Intercultural Adaptation Inventory consists of 49 items and is 6-point Likert type. A high score from the inventory indicates cultural compatibility, and a low score indicates incompatibility with the culture. The inventory assesses individuals' levels of intercultural activity and their abilities regarding individual awareness against the characteristics of the culture they live in. These dimensions are emotional flexibility (18 items), flexibility/openness (15 items), perceptual sensitivity (10 items), and personal autonomy (7 items). The Cronbach alpha internal consistency coefficient of the Intercultural Adaptation Inventory is 0.84.
THE PSYCHOLOGICAL WELL-BEING SCALE (PWS) | Change from before education up to after education (three weeks)
  The scale developed by Diener et al. (2010) was developed to measure socio-psychological well-being, complementing existing well-being measures. The Turkish adaptation of the scale was carried out by Telef in 2013. The Single Factor Psychological Well-Being Scale consists of 8 items and is in 7-point Likert type. All items are expressed positively. Scores from the scale range from 8 to 56. The higher the score obtained from the scale, the higher the level of psychological well-being is calculated. The Cronbach alpha internal consistency coefficient of the scale is 0.80.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal ALTUNDAL DURU, Doctor, Study Chair — Çankırı Karatekin University
Locations (1):
- Hilal ALTUNDAL DURU, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No